CLINICAL TRIAL: NCT07024550
Title: Evaluation of Changes in Brain Reward Pathway Activity After rTMS Therapy Via fMRI (Functional Magnetic Resonance Imaging)
Brief Title: Impact of the EXOMIND (BTL-699-2) on the Brain Reward Pathway
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-699_CTCZ200
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Binge Eating Behaviour; Binge Eating/Loss of Control Eating; Food Craving
Keywords: brain reward pathway; fMRI; brain activity; rTMS; ExoTMS; EXOMIND
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with BTL-699-2 device (Experimental): During six treatments, the subjects will be exposed to the electromagnetic field delivered non-invasively by the BTL-699-AP M-2 applicator placed on the left dlPFC.
  Interventions: Device: Treatment with BTL-699-2 device
- Treatment with BTL-699-2 device with intensity below therapeutic threshold (Sham Comparator): During six treatments, the subjects will be exposed to the electromagnetic field delivered non-invasively by the BTL-699-AP M-2 applicator placed on the left dlPFC, with the intensity of the energy set below the therapeutic threshold.
  Interventions: Device: Treatment with BTL-699-2 device with intensity below therapeutic threshold

INTERVENTIONS:
Device: Treatment with BTL-699-2 device — The treatment schedule with BTL-699-2 device will consist of six 24.5-minute treatments spaced 3-7 days apart. The therapy parameters will be adjusted according to patient feedback, but should never exceed 70% of the individual's MT in the active group.
  Other Names: Treatment with EXOMIND (BTL-699-2) device
  Arms: Treatment with BTL-699-2 device
Device: Treatment with BTL-699-2 device with intensity below therapeutic threshold — The treatment schedule with BTL-699-2 device will consist of six 24.5-minute treatments spaced 3-7 days apart. The intensity of the energy will be set below the therapeutic threshold.
  Other Names: Treatment with EXOMIND (BTL-699-2) device with intensity below therapeutic threshold
  Arms: Treatment with BTL-699-2 device with intensity below therapeutic threshold

SUMMARY:
The goal of this clinical trial is to thoroughly explore and ascertain the mechanism of action of the therapy with the EXOMIND (BTL-699-2) device in the treatment of food cravings (serving as an important precipitant to binge eating episodes), among binge eaters and to confirm its efficacy and safety, in adult binge-eating patients with food cravings. The main question it aims to answer is:

To ascertain the mechanism of action of the treatment with the EXOMIND (BTL-699-2) device equipped with a BTL-699-AP-M-2 applicator in reducing food cravings, for the active group only.

Participants will complete six treatments and one follow-up visit.

DETAILED DESCRIPTION:
The study is a prospective, single-center, two-arm, randomized controlled trial.

The subjects will be enrolled and randomly assigned to an active or sham experimental study arm. The ratio of active:sham groups will be 3:1.

The subjects will be required to complete six (6) treatment visits and one (1) follow-up visit, scheduled 1 month post-treatment.

At the screening visit, an informed consent will be obtained from the patient, and inclusion and exclusion criteria will be verified. A thorough medical history, review of concomitant medications and psychiatric examination will be performed, mainly focused on possible contraindications, to exclude subjects with a possible confounding condition. A drug and pregnancy test will be performed as part of the exclusion criteria assessment. Additionally, as a part of the inclusion criteria, subjects will be asked to fill out the Food Craving Questionnaire-Trait (FCQ-T) to evaluate the severity of the food cravings. The subject's motor threshold (MT) will be established as a part of the inclusion criteria.

Only subjects meeting all inclusion and none of the exclusion criteria will be enrolled, randomized (to a sham or active study group) and invited to baseline visit no later than 14 days after the screening visit. Baseline measurements will include recording the subject's weight and height to calculate their BMI (Body Mass Index). The performed MRI (Magnetic Resonance Imaging) scanning will be divided into collecting structural MRI and fMRI (during the food-cue reactivity task) to obtain pre-treatment data for subsequent analysis. During the baseline fMRI food-cue reactivity task measurement, the EEG (Electroencephalography) of the patients will be also collected.

The treatment administration phase consists of six (6) 24.5-minute treatment visits scheduled 3-7 days apart. After all pre-treatment procedures are completed, the first study treatment can be administered during the baseline visit. The BTL-699-AP-M-2 applicator will be positioned to cover the left dlPFC (Dorsolateral Prefrontal Cortex). The therapy parameters will be adjusted according to patient feedback, but should never exceed 70% of the individual's MT in the active group. The sham group will be treated with a 5% intensity of the individual's MT. The treatment area will be examined for possible adverse events after each treatment. After the last treatment, review of concomitant medications will be performed, the subjects will be weighed, asked to undergo pregnancy test, fMRI and fill out the FCQ-T, Subject Satisfaction Questionnaire (SSQ), and Therapy Comfort Questionnaire (TCQ). Structural MRI scans will also be collected before the fMRI scanning to detect any potential abnormalities in the treated area. Additionally, the EEG of the patients will be also collected in the course of the fMRI food-cue reactivity task. Before and after each treatment visit, and at the follow-up visit, an examination for possible adverse effects will be done.

The follow-up visit will be scheduled 1 month after the last treatment (±5 days). Review of concomitant medications will be performed, subjects will be weighed and asked to undergo pregnancy test, fMRI, to complete the Subject Satisfaction Questionnaire and FCQ-T. Structural MRI scans will also be collected before the fMRI scanning to detect any potential abnormalities in the treated area. Additionally, the EEG of the patients will be also collected in the course of the fMRI food-cue reactivity task.

The study outcomes will be based on exploring the differences in the neural activity post vs. pre-treatment in the active group and comparing the assessments' results of the active group to the sham group.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years
* Any self-reported excessive overeating episodes in the last 2 months
* The minimal pre-treatment FCQ-T score of 100 points
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb at least five out of ten times
* Subjects willing and able to abstain from partaking in any other weight management procedures (including diet and exercise regime changes) other than the study procedure during the study participation
* Subjects willing and able to abstain from initiating any other eating disorder treatments other than the study procedure during the study participation
* Subjects willing and able to undergo fMRI scanning, structural MRI scanning, and EEG recording, and proceed with the instructions from the study staff during the measurement
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* If applicable, subjects will maintain pre-study prescribed medications at a stable therapeutic dosage and/or with maintained frequency of psychotherapy during the study participation. The pre-study treatment regime needs to be set and maintained for at least 2 months prior to the study enrollment

Exclusion Criteria:

* Electronic implants (Implanted stimulator devices in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants including device leads, deep brain stimulators, cochlear implants, ocular implants, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, and neurostimulator.)
* metallic, ferromagnetic or other magnetic-sensitive implants/objects in or near the head - rTMS devices are contraindicated for use in patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head (with some exceptions in the mouth - see the Safety Precautions and Warnings) or within 30 cm of the treatment coil. (Examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewellery, and hair barrettes).
* application in the heart area
* persons with a tendency to seizure (hypotonic, epileptic)
* ongoing anticoagulation therapy
* ongoing severe or life-threatening condition
* ongoing renal dialysis therapy or decompensated renal insufficiency
* decompensated hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases
* malignant or benign tumour (within 30 cm of the treatment coil)
* fever
* application over or in the near proximity (within 30 cm of the treatment coil) of tattoos with metallic ink
* Shrapnel or other metal or electronic implants (pacemakers, surgical devices, metallic tattoos on the head, etc.)
* pregnancy or lactation, absence of medically approved contraceptive methods in females of childbearing potential
* history of head trauma, increased intracranial pressure or fainting
* major medical, neurological, or psychological disorders (e.g. depression, panic attacks, ADHD, tumors, heart conditions, claustrophobia)
* current usage of sleeping aids, painkillers (including aspirin), or other agents known to affect brain function (e.g. antihistamines, decongestants)
* any other contraindications for MRI examination
* intake of one or a combination of the following drugs forms a strong potential hazard for the application of rTMS due to their significant seizure threshold-lowering potential: imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines (MDMA, ecstasy), cocaine, phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline
* intake of seizure threshold-lowering drugs such as mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, sympathomimetics
* withdrawal from one of the following drugs could form a relative hazard for the application of rTMS due to the resulting significant seizure threshold lowering potential: alcohol, barbiturates, benzodiazepines, meprobamate, chloralhydrate
* suicidal tendencies or recent attempt to commit suicide
* concurrent use of electroconvulsive therapy or vagus nerve stimulation
* other intake disorders such as bulimia, anorexia
* vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
* systemic infection
* patients with a broad of neuropsychiatric diseases are at elevated risk for seizures. Essentially all neurologic conditions with structural cerebral damage (e.g. stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers) are associated with an elevated risk for seizures
* immunosuppressive therapy with tacrolimus, and other agents which can cause the posterior reversible leukoencephalopathy syndrome
* diagnosis of post-traumatic stress disorder, psychotic disorder or current psychotic symptoms, bipolar disorder, borderline personality disorder
* pulmonary insufficiency
* heart disorders
* personal history of syncope (except the reflex syncope)
* implanted infusion pumps, drug pumps (within 30 cm of the treatment coil)
* contradictions for the testing used in the trial, for example, the motor threshold cannot be found or quantified
* any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in the brain reward pathway activity | baseline to 1 month post-treatment
  The treatment-induced changes in the reward pathway activity of the investigated brain regions detected via fMRI during the food-cue reactivity task for the participants in the active group.

SECONDARY OUTCOMES:
Assessment of changes in the FCQ-T (Food cravings questionnaire-trait) score for the active group vs. sham group at 1 month | baseline and 1 month post-treatment
  The change from the pre-treatment FCQ-T score in the active group compared to the sham group at the 1-month follow-up visit; score range (39-234), score reduction indicates reduction of food cravings
Subject satisfaction as assessed by Subject Satisfaction Questionnaire | baseline to 1 month post-treatment
  Evaluation of satisfaction of the treated subjects with the therapy based on the Subject Satisfaction Questionnaire; the ranking is based on the 5-point Likert scale (1-5), higher score means higher satisfaction
Comfort as assessed by Therapy Comfort Questionnaire | from the first to the last treatment session, assessed up to 42 days
  Evaluation of comfort of the treated subjects during the therapy based on the Therapy Comfort Questionnaire; the ranking is based on the 5-point Likert scale (1-5), higher score means higher comfort, and on the Numerical Analog scale (0-10), higher score means higher pain

OTHER OUTCOMES:
Incidence of Treatment-related Adverse Events | baseline to 1 month post-treatment
  The evaluation of the safety of the BTL-699-2 device through the occurrence of adverse effects and examination of the structural MRI scans.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health in Czechia, Klecany, Czechia